CLINICAL TRIAL: NCT05984823
Title: Home-based Body Weight Exercise With Blood Flow Restriction (BFR): Feasibility of a Novel Rehabilitation Intervention in COPD Patients
Brief Title: Home-based Body Weight Exercise With Blood Flow Restriction (BFR): Feasibility of a Novel Rehabilitation Intervention in COPD Patients (HomeBFR-COPD)
Acronym: HomeBFR-COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment target was less than the target due to the reduced time available within the researchers PhD timeline (funded registration period was 1st January 2022 to 31st December 2024)
Sponsor: Mrs Hanoof Aljohani (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor-Investigator, Mrs Hanoof Aljohani, Lead Investigator, Loughborough University
Organization: Loughborough University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HomeBFR-COPD
Record Dates: First submitted 2023-07-13; First posted 2023-08-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Blood flow restriction; Home-based exercise; Tele-health; Body weight strength exercise; Feasibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Intervention group and control group
Who Masked: Outcomes Assessor
Masking Description: The lead researcher performed baseline assessments prior to randomisation and was therefore blinded to group allocation. Participants were then randomised (1:1) by an independent researcher using a computer-generated sequence. Follow-up assessments were conducted by the same researcher, who was not blinded at that stage due to involvement in intervention delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Body weight exercise with blood flow restriction
  Interventions: Other: Home based body weight type exercises with blood flow restriction
- Exercise only group (Active Comparator): Body weight exercise only
  Interventions: Other: Home based body weight type exercises

INTERVENTIONS:
Other: Home based body weight type exercises with blood flow restriction — The participant will be asked to complete blood flow restricted exercises described below three times per week for 6 weeks.
  Exercise protocol: Two tourniquets will be placed around the upper part of each thigh, these tourniquets will be inflated to an individualised and maintained for the duration of each exercise (including the inter-set rest period) but deflated during the 5 min rest in between. Five Body weight Exercises will be performed: Sitting knee extensions, standing knee raise, Heel-toe raises, Bilateral, mini-squat behind a chair, and Chair rise/sit to stand.
  Arms: Intervention group
Other: Home based body weight type exercises — The participant will be asked to complete body weight exercises for three times per week for 6 weeks. These exercises include: Sitting knee extensions, standing knee raise, Heel-toe raises, Bilateral, mini-squat behind a chair, and Chair rise/sit to stand.
  Arms: Exercise only group

SUMMARY:
The primary aim of this randomised controlled trial is to investigate the feasibility and acceptability of low-intensity exercise with blood flow restriction (BFR) in patients with Chronic Obstructive Pulmonary disease (COPD).

The investigators will also collect functional and physiological outcome data to explore potential mechanisms and provide data for a power calculation to be used in a future randomised controlled trial (RCT) to ensure that subsequent full scale clinical RCT has maximum reach and benefit.

The primary experimental hypothesis that underpins these aims is:

• Low-intensity exercise with BFR is a tolerable, acceptable, and safe exercise modality in COPD patients.

40 patients attending clinics at University Hospitals of Leicester (UHL) National Health Service (NHS) Trust with diagnosed COPD will be randomly allocated to a home-based body weight exercise intervention either with or without the blood flow restriction (n=20 in each group). The body weight exercise will consist of five body weight exercises including: sitting knee extensions, standing knee raise, heel-toe raises, bilateral mini-squat behind a chair, and chair rise/sit to stand.

In addition to the pre and post intervention visits, the initial two training sessions for both groups will be directly supervised in the research centre. These sessions are to ensure all exercises are performed correctly and safely and the patient become familiar with the exercises and BFR equipment and mobile application, which provides exercise guidance and session recording.

DETAILED DESCRIPTION:
Experimental design:

This is a randomised, controlled, assessor blind, single centre, clinical trial. Outcome measurements will be assessed at baseline and following the 6-week home-based intervention.

Participants:

40 Eligible participants will be identified and approached by their own clinical team at routine clinical appointments or at the point of referral to pulmonary rehabilitation (PR). In addition, potential participants who didn't attend PR or are on the waiting list and individuals who have previously provided written consent to be contacted about future research studies will be contacted via post. If interested, a researcher will explain the study and provide the Participant Information Sheet. All participants will be given at least 48 hours to consider taking part and written informed consent will be obtained before any study procedure.

Experimental protocol:

Patients will be randomised (1:1 intervention: control ratio) matched for age and lung function to a home-based body weight exercise intervention including sitting knee extensions, standing knee raise, heel-toe raises, bilateral mini-squat behind a chair, and chair rise/sit to stand either with or without the blood flow restriction (n=20 in each group).

Baseline outcome measures will be conducted over the first visits to the clinic.

Initial two training sessions will be directly supervised in the research centre (visits 2 & 3) to ensure all exercises are performed correctly and safely and the patient become familiar with the trial equipment and related mobile application for exercise guidance and session recording (digital training). During both sessions, physiological measurements will be made frequently venous blood samples to assess markers of inflammation, immune and vascular health will be obtained. A brief survey to assess exercise experience will e completed at the end of visit 3.

Patients will then be asked to carry on by performing the same exercises three times per week at home for the next five weeks. The programme will start at a quite easy level and gradually increase in intensity every two weeks depending on how the participant gets on. Progression will incorporate an increase in the number of repetitions and sets every two weeks.

After the intervention phase, patients will return to the research centre for post-intervention assessment visit (visit 4) where post-intervention outcome measures (including a post-training resting blood sample) will be conducted over the same time-course as the baseline measures. at the end of the visit, a brief survey to assess exercise experience will be completed. In addition, half of the participants will be interviewed, within four weeks of completion of the study, to qualitatively assess perceived expectations, benefits, motives, and barriers to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged 40 years or above
* Diagnosed with COPD as per GOLD criteria (Forced expiratory volume(FEV1)/forced vital capacity(FVC) <0.7)
* FEV1 ≤ 80% predicted
* Medical Research Council (MRC) dyspnoea scale ≥2
* BMI <= 35
* Willing and able to give informed consent for participation in the study.
* Stable dose of current regular medication for at least 4 weeks prior to study entry.
* Clinically acceptable ECG at enrolment.
* Able (in the investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Unable to communicate sufficiently in English
* Unable to give informed consent or comply with testing and training protocol for any reason.
* Acute exacerbation in the preceding 4 weeks (would become eligible 4 weeks following recovery).
* Unable to undertake exercise due to physical or psychological barriers.
* Contraindication to exercise training (American College of Sports Medicine guidelines)
* Any major or uncontrolled comorbidity that would impair the participant's ability to exercise or would mean exercise was unsafe (e.g., uncontrolled diabetes, hypertension BP>160/100, muscle or joint injuries which would limit ability to exercise).
* Any other significant disease, disorder, or medical condition which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study including (but not limited to):

Any clotting disorder Any bleeding disorder (e.g., haemophilia) Recent (<3 months) venous thromboembolism, vascular (artery or vein) surgery to the legs, skin graft to the legs, and or arteriovenous fistula in the legs.

Had one or both legs immobilisation in the last 4 weeks (e.g., prolonged bed rest, or recent orthopaedic intervention) Taking any anticoagulant medication Significant peripheral neuropathy

* Current or within the last 3 months (or maximum relevant wash out period, whichever is longer), participation in an investigational medicinal product (IMP) or device trial at the time of screening.
* Current or within the last 6 months (or maximum relevant wash out period, whichever is longer), participation in pulmonary rehabilitation or in another research study involving exercise training.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Female participants who are pregnant, lactating, or planning pregnancy during the course of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rates | Through study completion, an average of 18 months
  The investigators estimate a recruitment rate of 15% with 95% Confidence interval of ± 7%. A recruitment rate of 15% is in line with the referral rate for PR in stable and post-exacerbation COPD.
Retention rates | Through study completion, an average of 18 months
  The investigators estimate a retention rate of 80% ± 19%. A retention rate of 80% is close to that seen in pre-pandemic PR programmes locally and is similar to that seen in our previous exercise studies.
Adherence to the intervention (in supervised and unsupervised sessions) | Through study completion, an average of 18 months
  The investigators estimate that individuals would complete a mean of 14 out of 18 training sessions (78%, 95% Confidence interval ± 10%).
Safety (adverse events) | Through study completion, an average of 18 months
  The investigators will monitor for potential adverse events that may be related to the intervention (venous thromboembolism, rhabdomyolysis, accelerated hypertension, altered lower limb sensation, localised bruising, clotting disorder) through specific screening questionnaires and blood pressure monitoring at study visits. Concerns about possible adverse events will result in direct referral to NHS services for further investigation and involvement in the study will be paused until these investigations have been completed.
Exercise experience | Through study completion, an average of 18 months
  Brief survey upon completion of supervised training sessions and upon completion of the study. Survey items build on previous research and relate to exercise experience.
Acceptability | Through study completion, an average of 18 months
  Qualitatively with in-depth, semi-structured, one-to-one exit interviews of 50% of participants (randomly chosen) 1 - 4 weeks after completion of the final follow-up assessment.Topics will focus on patients' perceived expectations, benefits, motives, and barriers to the intervention.
  - Examining reasons for declining to participate amongst eligible patients, reasons for non-adherence to the exercise intervention, and reasons for dropout amongst discontinuing patients.

SECONDARY OUTCOMES:
Aerobic exercise capacity (VO2peak) | At baseline visit (week 0) and follow up visit (week 7).
  VO2peak (ml/kg/min), will be assessed using an incremental-cycle-exercise test on a cycle ergometer which has a high precision for VO2peak confirmation and is well tolerated by patients.
Lower limb function | At baseline visit (week 0) and follow up visit (week 7).
  Short Physical Performance Battery (SPPB) will be performed consisting of tests of gait speed, standing balance, and chair stand tests. The SPPB consists of 3 individual sub-tests - standing balance, 4-meter gait speed (4mGS) and 5-repetition sit-to-stand (5STS).
Quadriceps muscles strength | At baseline visit (week 0) and follow up visit (week 7).
  Maximal isometric and isokinetic quadriceps strength of both legs using an isokinetic dynamometer.
Chronic Respiratory Questionnaire (CRQ) | At baseline visit (week 0) and follow up visit (week 7).
  A valuable health related quality of life (HRQL) tool that it incorporates patient perceptions of both physical and emotional health. Four aspects of HRQL are evaluated: dyspnoea, fatigue, emotional function, and mastery. Each domain includes 4 to 7 items, with each item graded on 7-point Likert scale; item scores within a domain are summated to provide a total score for each domain. Higher scores indicate better HRQL.
COPD Assessment Tool (CAT) | At baseline visit (week 0) and follow up visit (week 7).
  CAT questionnaire consists of eight items on a 1-to-5-point scale assessing various manifestations of COPD. It provides a simple quantified measure of health related quality of life (HRQL) focusing on cough, phlegm, chest tightness, breathlessness, limited activities, and confidence leaving home, sleeplessness, and energy. The total score is correlated with the impact level of COPD on health status and is interpreted as low (<10), medium (10-20), high (21-30) and very high (>30).
Hemodynamic response to exercise | At visit 2 and 3 (week 1) of supervised training sessions.
  Heart rate (beats per minute) will be monitored throughout exercise using chest strap heart rate sensor (Polar H10)
Hemodynamic response to exercise | At visit 2 and 3 (week 1) of supervised training sessions.
  Systolic and diastolic blood pressure (millimetres of mercury) will be continuously assessed during exercise using an ambulatory blood pressure monitor (The Oscar 2™)
Hemodynamic response to exercise | At visit 2 and 3 (week 1) of supervised training sessions.
  Oxygen saturations (%O2sat) will be monitored throughout exercise using Nonin 3150 WristOx2 Pulse Oximeter.
Muscle soreness | At visit 2 and 3 (week 1) of supervised training sessions.
  Muscle soreness will be assessed using a visual analog scale. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no soreness" and "extreme soreness".
Exercise intensity | At visit 2 and 3 (week 1) of supervised training sessions.
  Rate of perceived exertion will be continuously assessed during exercise using Modified Borg Dyspnoea Scale which uses a scale from 0 to 10, where 0 represents no dyspnea and 10 represents maximal dyspnea.
Concentration of skeletal muscle damage biomarker (CK) | Before, 1 hour after, and 48 hours after exercise at visit 2 of supervised training session (week 1) and at baseline of visit 4 (week 7).
  Venous blood samples will be obtained for measurement of skeletal muscle damage biomarker (CK).
Concentration of inflammation biomarkers including, CRP, interleukin-6, immune and endothelial cell-expressed soluble adhesion molecules. | Before, 1 hour after, and 48 hours after exercise at visit 2 of supervised training session (week 1) and at baseline of visit 4 (week 7).
  Venous blood samples will be obtained for measurement of inflammation biomarkers (CRP, interleukin-6, immune and endothelial cell-expressed soluble adhesion molecules).
Concentration of endothelial function biomarker (bradykinin). | Before, 1 hour after, and 48 hours after exercise at visit 2 of supervised training session (week 1) and at baseline of visit 4 (week 7).
  Venous blood samples will be obtained for measurement of endothelial function biomarker (bradykinin).
Concentration of cardiac cell injury and stretch biomarkers troponin I and BNP | Before, 1 hour after, and 48 hours after exercise at visit 2 of supervised training session (week 1) and at baseline of visit 4 (week 7).
  Venous blood samples will be obtained for measurement of cardiac cell injury and stretch biomarkers (troponin I and BNP).
The presence of endothelial progenitor cells | Before, 1 hour after, and 48 hours after exercise at visit 2 of supervised training session (week 1) and at baseline of visit 4 (week 7).
  Venous blood samples will be obtained for measurement of the presence of endothelial progenitor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ward, MBBS, PhD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- NIHR Leicester Biomedical Research Centre - Respiratory, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of research chief investigator and/or principal investigator.

REFERENCES:
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Clarkson MJ, Conway L, Warmington SA. Blood flow restriction walking and physical function in older adults: A randomized control trial. J Sci Med Sport. 2017 Dec;20(12):1041-1046. doi: 10.1016/j.jsams.2017.04.012. Epub 2017 Apr 21. PMID 28483555
- [Background] Patterson SD, Hughes L, Head P, Warmington S, Brandner C. Blood flow restriction training: a novel approach to augment clinical rehabilitation: how to do it. Br J Sports Med. 2017 Dec;51(23):1648-1649. doi: 10.1136/bjsports-2017-097738. Epub 2017 Jun 22. No abstract available. PMID 28642225
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Pereira-Neto EA, Johnston KN, Lewthwaite H, Boyle T, Fon A, Williams MT. Title: Blood flow restricted exercise training: Perspectives of people with chronic obstructive pulmonary disease and health professionals. Chron Respir Dis. 2021 Jan-Dec;18:14799731211056092. doi: 10.1177/14799731211056092. PMID 34823382
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Swallow EB, Reyes D, Hopkinson NS, Man WD, Porcher R, Cetti EJ, Moore AJ, Moxham J, Polkey MI. Quadriceps strength predicts mortality in patients with moderate to severe chronic obstructive pulmonary disease. Thorax. 2007 Feb;62(2):115-20. doi: 10.1136/thx.2006.062026. Epub 2006 Nov 7. PMID 17090575
- [Background] Madarame H, Kurano M, Fukumura K, Fukuda T, Nakajima T. Haemostatic and inflammatory responses to blood flow-restricted exercise in patients with ischaemic heart disease: a pilot study. Clin Physiol Funct Imaging. 2013 Jan;33(1):11-7. doi: 10.1111/j.1475-097X.2012.01158.x. Epub 2012 Jul 30. PMID 23216760